CLINICAL TRIAL: NCT01986413
Title: German: Einfluss Von Gesichertem Atemminutenvolumen Auf Schlafqualität Und Häufigkeit Respiratorischer Ereignisse Bei Patienten Mit Nicht Invasiver Beatmung (NIV)
Brief Title: Intelligent Volume Assured Pressure Support to Improve Sleep Quality and Respiratory Events in Patients With Non Invasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Georg Nilius, PD Dr. med., Helios Klinik Ambrock
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IVAPSleep 2013
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: COPD; Chronic Hypercapnic Respiratory Failure
Keywords: COPD; chronic hypercapnic respiratory failure; NIV; respiratory events; IVAPS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIPAP ST (Active Comparator): one night, NIV with pressure controlled ventilation (BIPAP ST) with individually titrated pressure parameters.
  Interventions: Device: pressure controlled ventilation BIPAP ST; Device: NIV
- IVAPS (Experimental): one night, NIV with volume assured pressure support (IVAPS).The pressure parameters will be adjusted according to the BIPAP pressure levels.
  Interventions: Device: volume assured pressure support IVAPS; Device: NIV

INTERVENTIONS:
Device: pressure controlled ventilation BIPAP ST — spontaneous timed pressure controled bilevel ventilation
  Other Names: Stellar™ 150, ResMed
  Arms: BIPAP ST
Device: volume assured pressure support IVAPS — intelligent volume assured Pressure Support
  Other Names: Stellar™ 150 with iVAPS
  Arms: IVAPS
Device: NIV — Patients with COPD and chronic hypercapnic respiratory failure will spent two nights on NIV, one with spontaneous timed pressure controlled bilevel ventilation (BiPAP ST) and one with the advanced mode of intelligent volume assured pressure support (IVAPS). Patients will spend the treatment nights in randomized order under polysomnographic surveillance, including transcutaneous PCO2 measurement.
  Other Names: Stellar™ 150, ResMed

SUMMARY:
Aim of this prospective randomized trial is to compare non invasive ventilation (NIV) with pressure control (BiPAP-ST) to volume assured pressure support (iVAPS) with regards to sleep quality and alveolar ventilation in patients with routine NIV initiation after COPD exacerbation.

20 patients with COPD and chronic hypercapnic respiratory failure will spent two nights on NIV, one with spontaneous timed pressure controlled bilevel ventilation (BiPAP-ST) and one with the advanced mode of intelligent volume assured pressure support (iVAPS). Patients will spend the treatment nights in randomized order under polysomnographic surveillance, including transcutaneous PCO2 measurement. Besides the number of arousals and PCO2 values over night the sleep quality will be judged with regards to especially adjusted respiratory event criteria like unintentional leaks, patient ventilator asynchrony, and decrease of ventilatory drive.

DETAILED DESCRIPTION:
Non invasive ventilation (NIV) is one of the major medical innovations of the last 30 years. Especially continuous positive airway pressure (CPAP) is the established Gold Standard in obstructive sleep apnea (OSA) treatment.

NIV with bilevel ventilation (BiPAP-ST) is the established Gold Standard in acute hypercapnic respiratory failure, especially in exacerbated COPD.

Still, the adaption of CPAP in OSA is less complicated than a bilevel therapy in hypercapnic failure. The adjustment of NIV requires not only the definition of expiration pressure (PEEP) but also of inspiration pressure support. Only adequate pressure difference guarantees effective ventilatory assistance and an improvement of alveolar ventilation. The pressure changes need to be defined by the physician, as well as the breathing frequency.

Ventilation can furthermore be controlled by a target volume (volume controlled) or a target pressure (pressure controlled).

Moreover, patients with respiratory insufficiency are often suffering of significant dyspnoea and are hard to accustom to a respiratory mask.

There is a lack of systematic studies addressing the effects of different ventilator settings on sleep and life quality, as well as studies about the necessary monitoring extent during the NIV initiation.

ELIGIBILITY:
Inclusion Criteria:

* Stable respiratory insufficiency
* Hypercapnia >50 mmHG
* Clinically required NIV
* Capable of giving consent

Exclusion Criteria:

* Existing ventilatory support
* Invasive ventilation
* Any other severe physical disease that requires immediate medical assistance
* Acute hypercapnic decompensation with pH <7.30 in routine BGA
* Circumstances that doesn't allow mask ventilation (e.g. facial deformation)
* Participation in a clinical trial within the last 4 weeks
* Pregnancy or nursing period
* Drug addiction

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of respiratory events during non invasive ventilation | 2 nights
  Unintentional leak, patient ventilator asynchrony, decrease of ventilatory drive, Apnoea, Hypopnea

SECONDARY OUTCOMES:
Sleep efficiency | 2 nights
  Relation between "time in bed" and "total sleep time" measured by a polysomnography under non invasive ventilation.

OTHER OUTCOMES:
mean PCO2-level during non invasive ventilation | 2 nights
  Mean pCO2 level over night measured transcutaneously with a polysomnography under non invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Helios Klinik Hagen
Locations (1):
- Helios Klinik Hagen, Hagen, North Rhine-Westphalia, Germany